CLINICAL TRIAL: NCT02793063
Title: Rare Diseases Clinical Research Network Brittle Bone Disorders Consortium Osteogenesis Imperfecta (OI) Quality of Life Survey Pilot Project 2
Brief Title: Osteogenesis Imperfecta (OI) Quality of Life Survey Pilot Project 2
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: BBD7702; U01TR001263 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2017-03

CONDITIONS: Osteogenesis Imperfecta; Brittle Bone Disorders
Keywords: Brittle Bone; Osteogenesis Imperfecta; BBD; OI; Congenital Abnormalities; Congenital Bone Disorder; Lobstein Syndrome
MeSH Terms: conditions — Osteogenesis Imperfecta; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BBD Consortium Contact Registrants: Osteogenesis Imperfecta patients who have self-registered at the Brittle Bone Disorders Consortium (BBD) Consortium Contact Registry, a web-based contact registry developed and supported by the Data Management and Coordinating Center (DMCC) for the Rare Diseases Clinical Research Consortium (RDCRN), located at the University of South Florida.
  Interventions: Other: Web-based Survey

INTERVENTIONS:
Other: Web-based Survey — This study will occur online. Participants will be asked to complete multiple surveys one time. Participants may receive study reminder emails to complete surveys. Participants will be able to complete the surveys all at once or in multiple sessions. Participants will have approximately 3 months to complete the surveys after consenting.

SUMMARY:
The purpose of this study is to explore the patient perspective of disease burden in Osteogenesis Imperfecta (OI). Participants will complete a web-based survey of questions which are usually administered within the Patient-Reported Outcome Measurement Information System (PROMIS) and provide feedback regarding the appropriateness of the questions for someone with OI.

DETAILED DESCRIPTION:
Participants will be recruited through the RDCRN BBD Contact Registry. An email invitation will be sent to all RDCRN BBD Contact Registry participants that meet the inclusion criteria to complete the online PROMIS CAT instruments. The email invitation will contain a link to the informed consent form. Once participants have consented to the study, they will have access to the online instruments. Follow-up emails will be sent to participants that have not completed any of the instruments. Reminder emails will be sent to participants with partially completed instruments.

Data will be collected and stored by the RDCRN DMCC at USF.

Data from patients co-enrolled in the "Longitudinal Study of Osteogenesis Imperfecta" and the BBD RDCRN Contact Registry will be linked and compared. Additional disease specific information will be collected by the survey (e.g., information on OI type and diagnosis, height, number of fractures, concurrent medication use, utilization of any mobility aid, hearing aid, or other device that they may use.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the RDCRN BBD Contact Registry English speaking Age 2 to adult

Exclusion Criteria:

* Inability to provide informed consent Inability to complete instruments

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Osteogenesis Imperfecta who are enrolled in the RDCRN BBD Contact Registry
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

PRIMARY OUTCOMES:
Validated Computer Adaptive Testing (CAT) PROMIS instruments | 3 months
  An online assessment will be used to obtain responses for each instrument. Scores for each are norm-based with a mean of 50 and standard deviation of 10 based upon the general population. Calibration of the standard error (SE) surrounding the reported score is possible. Default setting of 0.30 will be used for standard error with the minimum number of questions per item of 4 and maximum number of questions 8, using the computer adapted testing structure of the PROMIS instruments. Lower maximum number than the default settings will be used to avoid too many questions being given to a respondent when they do not report a diminished quality of life on any dimension. With these settings, survey respondents will be administered an average of 4-5 items per instrument and the testing among patients with OI indicate that the whole assessment will typically take 15-30 minutes in most instances.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Krischer, Ph.D., Principal Investigator — University of South Florida; Laura Tosi, M.D., Principal Investigator — Children's National Research Institute; Jeffrey Krischer, Ph.D., Study Chair — University of South Florida; Laura Tois, M.D., Study Chair — Children's National Research Institute
Locations (1):
- University of South Florida, Health Informatics Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richesson RL, Young K, Lloyd J, Adams T, Guillette H, Malloy J, Krischer JP. An automated communication system in a Contact Registry for persons with rare diseases: tools for retaining potential clinical research participants. AMIA Annu Symp Proc. 2007 Oct 11:1094. PMID 18694191
- [Result] Richesson RL, Lee HS, Cuthbertson D, Lloyd J, Young K, Krischer JP. An automated communication system in a contact registry for persons with rare diseases: scalable tools for identifying and recruiting clinical research participants. Contemp Clin Trials. 2009 Jan;30(1):55-62. doi: 10.1016/j.cct.2008.09.002. Epub 2008 Sep 7. PMID 18804556